CLINICAL TRIAL: NCT05282719
Title: A Multi-center, Phase II, Single-arm Clinical Study of Venetoclax Combined With Azacytiside in the Treatment of Myelodysplastic/Myeloproliferative Neoplasms in Adults
Brief Title: Clinical Study of Venetoclax Combined With Azacytiside in the Treatment of Myelodysplastic/Myeloproliferative Neoplasms in Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Head of Hematology Laboratory, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MDS/MPN-01
Record Dates: First submitted 2022-02-21; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Myelodysplastic/Myeloproliferative Neoplasms; Adult
MeSH Terms: conditions — Myelodysplastic-Myeloproliferative Diseases | interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment regime (Experimental): On day 1 of each cycle, decitabine 75 mg/m2 will be given subcutaneously, and will continue for 5 days. Simultaneously the patient will start out with Venetoclax 100mg and progress to 400mg until the 14 day cycle is finished.
  Interventions: Drug: venetoclax combined with azacitidine

INTERVENTIONS:
Drug: venetoclax combined with azacitidine — On day 1 of each cycle, decitabine 75 mg/m2 will be given subcutaneously, and will continue for 5 days. Simultaneously the patient will start out with Venetoclax 100mg and progress to 400mg until the 14 day cycle is finished.
  Other Names: combination of venetoclax plus azacitidine

SUMMARY:
To explore the efficacy of venetoclax combined with azacytidine in Myelodysplastic / myeloproliferative neoplasms（MDS/MPN）, so as to improve the overall survival and treatment status of MDS/MPN patients.

DETAILED DESCRIPTION:
At present, there is no standardized treatment strategy for MDS/MPN. The purpose of our study is to explore the efficacy of venetoclax combined with azacytidine in the treatment of MDS/MPN, so as to improve the overall survival and treatment status of patients with MDS/MPN. After the participants were treated with four cycles of venetoclax combined with azacytidine, the efficacy was evaluated according to the 2015 adult MDS/MPN response criteria to determine the disease status. Participants with disease progression and intolerance withdrew from the study during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age (years) >= 18；
2. Patients newly diagnosed or previously treated with MDS/MPNs (CMML, MDS/MPN-U, aCML) according to 2016 WHO diagnostic criteria:

   Initial diagnosis: CMML: CPSS-mol intermediate risk 2 and above; aCML; MDS/MPN-U.

   Previous treatment: HMA treatment failed.
3. Eastern Cooperative Oncology Group (ECOG) Performance status of 0,1, 2 ;
4. Liver function: Total bilirubin ≤3 upper limit of normal (ULN); aspartate aminotransferase (AST) ≤3 ULN; alanine aminotransferase (ALT)≤3 ULN；
5. Renal function#Ccr ≥30 ml/min;
6. Patients who sign the informed consent must have the ability to understand and be willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Acute myeloid leukemia
2. Myelodysplastic syndrome
3. Subjects who had previously been treated with Venetoclax
4. Subjects who are known to be allergic to ingredients of the study drug or their analogues
5. HIV infection
6. HBV-DNA or HCV-RNA positive
7. Subjects with grade 2 or above cardiac failure and those considered unsuitable for inclusion by the investigator
8. Subjects who are pregnant or breastfeeding
9. Subjects reject to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Study start date to study end date, or death, whichever comes first, up to 4 years
  ORR (equals the rates of complete remission [CR]+partial remission [PR]+complete cytogenetic remission [CCyR]+marrow response [MR[+clinical benefit [CB] )of venetoclax in combination with azacitidine.
  1. CR and CCyR are shown in the secondary outcome measures below.
  2. PR: Normalization of peripheral counts and hepatosplenomegaly with bone marrow blasts (and blast equivalents) reduced by 50%, but remaining>5% of cellularity except in cases of MDS/MPN with≤5% bone marrow blasts at baseline.
  3. MR: Optimal marrow response: Presence of all marrow criteria necessary for CR without normalization of peripheral blood indices.
     Partial marrow response: Bone marrow blasts (and blast equivalents) reduced by 50%, but remaining>5% of cellularity, or reduction in grading of reticulin fibrosis from baseline on at least 2 bone marrow evaluations spaced at least 2 months apart.
  4. CB: Hematology improvement, spleen response and symptom response.

SECONDARY OUTCOMES:
Complete remission rate | Study start date to study end date, or death, whichever comes first, up to 4 years
  1. Bone marrow: ≤5% myeloblasts (including monocytic blast equivalent in case of CMML) with normal maturation of all cell lines and return to normal cellularity Osteomyelofibrosis absent or equal to "mild reticulin fibrosis" (≤grade 1 fibrosis).
  2. Peripheral blood: Leukocyte≤10×10E9 cells/L; Hemoglobin≥11g/dL; Platelets≥100×10E9/L, ≤450×10E9/L; Neutrophils≥1.0×10E9/L; Blasts 0%; Neutrophil precursors reduced to≤2%; Monocytes ≤1.0× 10E9/L.
  3. Extramedullary disease: Complete resolution of extramedullary disease present before therapy (eg, cutaneous disease, disease-related serous effusions), including palpable hepatosplenomegaly.
Complete remission rate of bone marrow morphology | Study start date to study end date, or death, whichever comes first, up to 4 years
  Presence of all marrow criteria necessary for CR without normalization of peripheral blood indices as presented above.
Hematology improvement (HI) rate | Study start date to study end date, or death, whichever comes first, up to 4 years
  Percentages of participants with HI (erythroid/platelet/neutrophil responses)
  1. Erythroid response: Hemoglobin increase by≥2.0 g/dL; Transfusion independence (TI) for ≥8 week for patients requiring at least 4 packed red blood cell transfusions in the previous 8 week; Only red blood cell transfusions given based on physician's judgment for a pretreatment Hgb of ≤8.5 g/dL will count in the red blood cell TI response evaluation.
  2. Platelet response: TI when previously requiring platelet transfusions of at least a rate of 4 platelet transfusions in the previous 8 week; Pretreatment≤20×10E9/L: increase from<20×10E9/L to>20×10E9/L and by at least 100%; Pretreatment>20×10E9/L but≤100×10E9/L: absolute increase of ≥30×10E9/L.
  3. Neutrophil response: Pretreatment≤0.5×10E9/L at least 100% increase and an absolute increase≥0.5×10E9/L; Pretreatment>0.5×10E9/L and≤1.0×10E9/L, at least 50% increase and an absolute increase ≥0.5×10E9/L.
Complete cytogenetic remission rate | Study start date to study end date, or death, whichever comes first, up to 4 years
  Resolution of previously present chromosomal abnormality (known to be associated with myelodysplastic, syndrome myeloproliferative neoplasms, or MDS/MPN), as seen on classic karyotyping with minimal of 20 metaphases or FISH.
Incidence of severe infection (≥grade 3 ) | Study start date to study end date, or death, whichever comes first, up to 4 years
  Assessed using CTCAE 5
Spleen response rate | Study start date to study end date, or death, whichever comes first, up to 4 years
  Either a minimum 50% reduction in palpable splenomegaly of a spleen that is at least 10 cm at baseline or a spleen that is palpable at more than 5 cm at baseline becomes not palpable.
Symptom response rate | Study start date to study end date, or death, whichever comes first, up to 4 years
  Improvement in symptoms as noted by decrease of ≥50% as per the MPN-SAF TSS scoring<20 were not considered eligible for measuring clinical benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, Professor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China